CLINICAL TRIAL: NCT07204990
Title: BELUGA: Better to Exchange ETT for LMA Before Extubation in Children Under General Anaesthesia
Acronym: BELUGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Telethon Kids Institute (Other)
Collaborators: Uppsala University Hospital (Other); Atrium Health Wake Forest Baptist (Other); Children's Hospital of Philadelphia (Other); Insel Gruppe AG, University Hospital Bern (Other); University of Sao Paulo (Other); Istituto Giannina Gaslini (Other); Child and Adolescent Health Service - Perth (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RGS0000007646
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Endotracheal Extubation; Airway Anesthesia; Paediatric
Keywords: Paediatrics; Anaesthesia; Surgery; Extubation; Respiratory adverse events

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ETT awake (Active Comparator): ETT removal once the patient is fully awake (at least 3 of the following criteria:
  spontaneous tidal volume >5ml/kg, conjugate gaze, facial grimace, eye-opening, purposeful movement)
  Interventions: Procedure: Endotracheal tube removed awake
- Group LMA exchange (Active Comparator): ETT removal deep; @ at least 1 Mac or an equivalent depth of anaesthesia (if available BIS<60, Sedline <50), an additional bolus of propofol (1mg/kg) maybe given if deemed appropriate/ required prior to the ETT removal. Following gentle suctioning around the ETT at the end of the case, the ETT is removed under deep anaesthesia and a LMA inserted.
  Interventions: Procedure: Laryngeal mask airway inserted following deep extubation

INTERVENTIONS:
Procedure: Endotracheal tube removed awake — Patient will have the ETT removed awake and transferred to PACU breathing independently or with a face mask.
  Arms: Group ETT awake
Procedure: Laryngeal mask airway inserted following deep extubation — Patient will have LMA inserted following deep extubation of endotracheal tube.
  Arms: Group LMA exchange

SUMMARY:
During surgery, anaesthetists can use an endotracheal tube (ETT) to facilitate ventilation. At emergence from general anaesthesia, there are two techniques for removal of the ETT: (1) the ETT is removed when the child is waking up in (awake removal); or (2) the ETT is removed while still under anaesthesia(deep removal).

Currently there is no evidence to suggest either technique is safer - deep removal of the ETT may decrease the risk of overall airway complications, including cough and desaturations. However, it may be associated with increased airway obstruction compared with awake extubation in paediatric patients. In our institution, a further technique has become increasingly common practice: removing ETT deep to avoid coughing and desaturation, then inserting a laryngeal mask airway (LMA) which can be removed once the patient is awake in the postoperative care unit (PACU), avoiding the risk of airway obstruction coupled with deep airway removal. The aim of the study is to assess whether deep removal of an ETT and exchange to an LMA, is superior to awake ETT removal with regards to the occurrence of postoperative respiratory adverse events.

In this study, patients will be randomised to awake removal of ETT or deep removal of an ETT and exchange to an LMA. Data will be collected regarding the rate of respiratory adverse events in either group, as well as the incidence of post-operative pain, delirium and nausea and vomiting.

DETAILED DESCRIPTION:
Anaesthesia induction and maintenance will be performed as deemed appropriate by the attending anaesthetist. The choice and dose of analgesia will be at the discretion of the individual anaesthetist adjusted to the individual patient's needs. All clinical care will be in accordance with institutional standards.

All children undergoing surgery under general anaesthesia involving insertion of an endotracheal tube who arrive in the PCH post-anaesthetic care unit (PACU) between 0800 and 1800 on weekdays during the data collection periods will be included in this study under a waiver of consent. Surgical lists in our institution operate on four-week cycles (weeks A, B, C and D), with some surgical specialities scheduled for one list a fortnight or one list every four weeks and others having multiple lists per week. In order to ensure that both intervention groups have equal representation of each of the weeks A, B C and D, data collection will take place in 8-week blocks until such a time as the sample size has been reached.

Group ETT awake: ETT removal once the patient is fully awake (at least 3 of the following criteria: spontaneous tidal volume >5ml/kg, conjugate gaze, facial grimace, eye-opening, purposeful movement Group LMA exchange: ETT removal deep; @ at least 1 Mac or an equivalent depth of anaesthesia (if available BIS <60, Sedline <50), an additional bolus of propofol (1mg/kg) maybe given if deemed appropriate/ required prior to the ETT removal as per normal clinical practice. Following gentle suctioning around the ETT at the end of the case, the ETT is removed under deep anaesthesia and a LMA is inserted in its place.

There is no individual randomisation or blinding in this study. Extubation procedure (either ETT removed awake or ETT removed deep and exchanged for LMA) will each be used for 4 out of 8 weeks during the data collection period. The intervention assigned for the first 4-week cycle of the data collection period will be decided by the toss of a coin. Thereafter, intervention 1 (either ETT awake or LMA exchange) will be in place for weeks 4 weeks, with the alternate intervention in place for the subsequent 4 weeks. Given the nature of the intervention it is not possible to have blinding for this study. The statistical analysis will be performed by individuals blinded to the randomisation. This will be repeated until the required sample size has been reached

Demographic information routinely collected as part of normal clinical care will be recorded on a patient data sheet, including their date of birth, natal sex, height, weight, ethnicity and age on the day of surgery. Details about their condition on the day of surgery will be collected, including their American Society of Anaesthesiologists physical status (ASA) I-IV, any upper respiratory tract infections in the last two weeks, current or previous respiratory risk factors, and any signs of obstructive sleep apnoea, details of know abnormal pulse oximetry, risk factors for postoperative nausea and vomiting and any history of prematurity. Details of their anaesthetic management and their time spend in the post-anaesthetic care unit (PACU) will also be recorded, as well as any incidence of respiratory adverse events at any time from induction of anaesthesia until discharge from PACU. Incidence of sore throat or hoarse voice will be collected on the day of surgery 2-4 hours post PACU discharge.

ELIGIBILITY:
Participant Inclusion Criteria

* Children 0-16 years,
* 5kg and above,
* presenting for elective, semi-elective or emergency surgery under general anaesthesia
* With airway management planned with an endotracheal tube.

Exclusion Criteria:

* Children with severe cardiopulmonary disease or syndrome
* Children < 5kg
* Children with a contraindication to deep removal of ETT deep or exchange of ETT to LMA at the end of the case (e.g. high risk of aspiration)
* Children with a known or anticipated difficult airway
* Children remaining intubated post-procedure
* Children undergoing major airway surgery or bronchoscopies

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2029-01-12 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Compare the overall rate of perioperative respiratory adverse events in children following either (1) awake removal of ETT or (2) exchange of ETT for LMA followed by awake removal of LMA | Assessed by the anaesthetist along the course of the patient's perioperative pathway from extubation until their discharge from the post-anaesthetic care unit (PACU)
  Perioperative respiratory adverse events (PRAE) are defined as:
  Major PRAE: laryngospasm or bronchospasm, as determined by the anaesthetist, or desaturation <85% SpO2 for more than 1 minute on pulse oximetry.
  Minor PRAE: desaturation (<85% SpO2 for more than 10 secs on pulse oximetry), airway obstruction, severe coughing, post-operative stridor.

SECONDARY OUTCOMES:
Compare the rate of specific perioperative respiratory adverse events in children following either (1) awake removal of ETT or (2) exchange of ETT for LMA followed by awake removal of LMA | Assessed by the anaesthetist along the course of the patient's perioperative pathway from extubation until their discharge from the post-anaesthetic care unit (PACU)
  Perioperative respiratory adverse events (PRAE) are defined as:
  Major PRAE: laryngospasm or bronchospasm, as determined by the anaesthetist, or desaturation <85% SpO2 for more than 1 minute on pulse oximetry.
  Minor PRAE: desaturation (<95% SpO2 for more than 10 seconds on pulse oximetry), airway obstruction, severe coughing, post-operative stridor.
  Each individual PRAE (laryngospasm, bronchospasm, desaturation, airway obstruction, severe persistent coughing and post-operative stridor) will be considered separately.
Compare the rate of required post-operative airway interventions in children following either (1) awake removal of ETT or (2) exchange of ETT for LMA followed by awake removal of LMA | Any airway interventions given along the course of the patient's perioperative pathway from extubation until their discharge from the post-anaesthetic care unit (PACU) will be recorded
  Airway interventions are defined as: requirement for jaw thrust after airway removal, CPAP, supplemental O2 for over 10 min after the airway has been removed awake, need to reinsert LMA or ETT, use of airway adjuncts (e.g. guedel once airway removed), need for propofol or muscle relaxant following airway removal.
Comparison of postoperative delirium scores in PACU (post anaesthetic care unit)between the two groups using the Paediatric Anaesthesia Emergence Delirium (PAED) scale 10 minutes after awake (UMSS <2) | A single measurement of using the PAED score will be taken 10 minutes after the patient is assessed to first be at a UMSS of 2 as per the PACU nurse.
  PAED scale ranges from 0 to 20, a score of 0 is equivalent to no delirium and 20 is significant delirium
Comparison of pain scores 5 and 20 min post-awake airway removal (ETT in the awake ETT group and LMA removal in the exchange group) between the two groups | Assessments of pain will be taken at 5 and 20 minutes after the patient is assessed to first be at a UMSS of 2 as per the PACU nurse.
  Pain will be assessed by the PACU nurse by asking the patient to rate their pain on a scale of 0 to 10, where 0 is no pain and 10 is worst possible pain.
Comparison of the number of additional opioid analgesia use in PACU between the two groups | All opioid analgesia usage from PACU admission until discharge will be recorded.
  Looking at the number of additional opioid analgesia patients need in each group and comparing these.
Comparison of time between the end of surgery and arrival in PACU between the two groups and time to UMSS <2 (awake) | Time at which patient arrives in PACU and time at which their UMSS score is ≤2 will be measured by the PACU nurse during their post-operative PACU admission. Measured in minutes/hours on day of surgery for each patient.
  End of surgery is defined as completed application of dressing/cast (as applicable). This will be minutes to hours of time.
Comparison of PACU time between the two groups | PACU time is defined as the time from arrival in PACU until ready for discharge from PACU.
To compare rates of vomiting and self-reported nausea in PACU between the two groups | Assessed from the time at which the patient is admitted to PACU until the time that they are discharged.
  Rates of vomiting will be as reported by the PACU nurse. Self-reported nausea will be recorded only in children over the age of 6 years.
To compare the incidence of sore throat and hoarse voice between the two groups | Collected on the day of surgery, 2-4 hours post discharge from PACU.
  Sore throat score as rated on a 4-point scale - nil, mild, moderate, severe. Hoarse voice as identified by parent and rated on a 4-point scale nil, mild, moderate, severe.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Australia (2):
  - Perth Children's Hospital, Nedlands, Western Australia
  - The Kids Research Institute Australia, Nedlands, Western Australia
- University of São Paulo, São Paulo, Brazil
- Istituto Giannina Gaslini, Genova, Italy
- Uppsala University Hospital, Uppsala, Sweden
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No